CLINICAL TRIAL: NCT05016882
Title: Efficacy and Safety Investigation of NNC0194-0499 Co-administered With Semaglutide in Subjects With Non-alcoholic Steatohepatitis: a Dose-ranging, Placebo Controlled Trial
Brief Title: Research Study on Whether a Combination of 2 Medicines (NNC0194 0499 and Semaglutide) Works in People With Non-alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9500-4656; U1111-1255-5551 (Other: World Health Organization (WHO)); 2020-003566-39 (EudraCT Number)
Record Dates: First submitted 2021-08-18; First posted 2021-08-23 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: This is a randomised, double-blind, active and placebo-controlled, double-dummy, parallel group, multinational trial investigating NNC0194-0499 at 3 different dose levels when co administered with semaglutide
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- NNC0194-0499 7.5 mg + semaglutide 2.4 mg (Experimental): Each subject will receive two subcutaneous injections once weekly, consisting of two active drugs or one active drug and one placebo or two placebo injections.
  Interventions: Drug: NNC0194 0499 50 mg/mL; Drug: Semaglutide 3 mg/mL
- Placebo (NNC0194-0499) 7.5 mg + semaglutide placebo 2.4 mg (Placebo Comparator): Each subject will receive two subcutaneous injections once weekly, consisting of two active drugs or one active drug and one placebo or two placebo injections.
  Interventions: Drug: Placebo (NNC0194-0499); Drug: Semaglutide placebo
- NNC0194-0499 15 mg + semaglutide 2.4 mg (Experimental): Each subject will receive two subcutaneous injections once weekly, consisting of two active drugs or one active drug and one placebo or two placebo injections.
  Interventions: Drug: NNC0194 0499 50 mg/mL; Drug: Semaglutide 3 mg/mL
- Placebo (NNC0194-0499) 15 mg + semaglutide placebo 2.4 mg (Placebo Comparator): Each subject will receive two subcutaneous injections once weekly, consisting of two active drugs or one active drug and one placebo or two placebo injections.
  Interventions: Drug: Placebo (NNC0194-0499); Drug: Semaglutide placebo
- NNC0194-0499 30 mg + semaglutide 2.4 mg (Experimental): Each subject will receive two subcutaneous injections once weekly, consisting of two active drugs or one active drug and one placebo or two placebo injections.
  Interventions: Drug: NNC0194 0499 50 mg/mL
- NNC0194-0499 30 mg + semaglutide placebo 2.4 mg (Experimental): Each subject will receive two subcutaneous injections once weekly, consisting of two active drugs or one active drug and one placebo or two placebo injections.
  Interventions: Drug: NNC0194 0499 50 mg/mL; Drug: Semaglutide placebo
- Placebo (NNC0194-0499) 30 mg + semaglutide 2.4 mg (Active Comparator): Each subject will receive two subcutaneous injections once weekly, consisting of two active drugs or one active drug and one placebo or two placebo injections.
  Interventions: Drug: Placebo (NNC0194-0499); Drug: Semaglutide 3 mg/mL
- Placebo (NNC0194-0499) 30 mg + semaglutide placebo 2.4 mg (Placebo Comparator): Each subject will receive two subcutaneous injections once weekly, consisting of two active drugs or one active drug and one placebo or two placebo injections.
  Interventions: Drug: Placebo (NNC0194-0499); Drug: Semaglutide placebo
- NNC0174-0833 2.4 mg + semaglutide 2.4 mg (Experimental): Each subject will receive two subcutaneous injections once weekly, consisting of two active drugs or one active drug and one placebo or two placebo injections.
  Interventions: Drug: Semaglutide 3 mg/mL; Drug: NNC0174 0833 10 mg/mL
- Placebo (NNC0174-0833) 2.4 mg + semaglutide placebo 2.4 mg (Placebo Comparator): Each subject will receive two subcutaneous injections once weekly, consisting of two active drugs or one active drug and one placebo or two placebo injections.
  Interventions: Drug: Semaglutide placebo; Drug: NNC0174 0833 placebo

INTERVENTIONS:
Drug: NNC0194 0499 50 mg/mL — Patients will receive subcutaneous (s.c., under the skin) injections of NNC0194-0499 once weekly The study will last for about 19 months
  Arms: NNC0194-0499 15 mg + semaglutide 2.4 mg; NNC0194-0499 30 mg + semaglutide 2.4 mg; NNC0194-0499 30 mg + semaglutide placebo 2.4 mg; NNC0194-0499 7.5 mg + semaglutide 2.4 mg
Drug: Placebo (NNC0194-0499) — Patients will receive subcutaneous (s.c., under the skin) injections of placebo once weekly The study will last for about 19 months
  Arms: Placebo (NNC0194-0499) 15 mg + semaglutide placebo 2.4 mg; Placebo (NNC0194-0499) 30 mg + semaglutide 2.4 mg; Placebo (NNC0194-0499) 30 mg + semaglutide placebo 2.4 mg; Placebo (NNC0194-0499) 7.5 mg + semaglutide placebo 2.4 mg
Drug: Semaglutide 3 mg/mL — Patients will receive subcutaneous (s.c., under the skin) injections of semaglutide once weekly The study will last for about 19 months
  Arms: NNC0174-0833 2.4 mg + semaglutide 2.4 mg; NNC0194-0499 15 mg + semaglutide 2.4 mg; NNC0194-0499 7.5 mg + semaglutide 2.4 mg; Placebo (NNC0194-0499) 30 mg + semaglutide 2.4 mg
Drug: Semaglutide placebo — Patients will receive subcutaneous (s.c., under the skin) injections of semaglutide placebo once weekly The study will last for about 19 months
  Arms: NNC0194-0499 30 mg + semaglutide placebo 2.4 mg; Placebo (NNC0174-0833) 2.4 mg + semaglutide placebo 2.4 mg; Placebo (NNC0194-0499) 15 mg + semaglutide placebo 2.4 mg; Placebo (NNC0194-0499) 30 mg + semaglutide placebo 2.4 mg; Placebo (NNC0194-0499) 7.5 mg + semaglutide placebo 2.4 mg
Drug: NNC0174 0833 10 mg/mL — Patients will receive subcutaneous (s.c., under the skin) injections of NNC0174-0833 once weekly The study will last for about 19 months
  Arms: NNC0174-0833 2.4 mg + semaglutide 2.4 mg
Drug: NNC0174 0833 placebo — Patients will receive subcutaneous (s.c., under the skin) injections of NNC0174-0833 placebo once weekly The study will last for about 19 months
  Arms: Placebo (NNC0174-0833) 2.4 mg + semaglutide placebo 2.4 mg

SUMMARY:
This study is being done to see if a combination of 2 medicines (called NNC0194-0499 and semaglutide) can reduce liver damage in patients with non alcoholic steatohepatitis (NASH).

NNC0194-0499 is a new medicine which works in the liver. Semaglutide is a well-known medicine, which is already used by doctors to treat type 2 diabetes in many countries. It also helps with weight loss and may reduce liver damage, and so prevent future liver complications. It works in a different way to NNC0194 0499. The 2 medicines may work better together than on their own.

The study will also look at a combination of semaglutide and another weight-loss medicine called NNC0174-0833, which may be another treatment option for NASH.

Each week, participants will get 2 injections. These could be 2 of the 3 medicines OR 1 of the medicines and a placebo OR 2 placebo injections. Which treatment participants get is decided by chance. A placebo is a dummy medicine which looks like the real medicine but doesn't contain any active medicine.

The study will last for about 19 months. Participants will have 14 clinic visits and 9 phone calls with the study doctor.

Participants will have 1 or 2 liver biopsies (tiny pieces of liver tissue) - one at the start (if participants have not had a biopsy recently) and one at the end of the study treatment.

Women: Women cannot take part if pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Aged greater than or equal to 18 years at the time of signing informed consent. In Republic of Korea, subjects must be aged greater than or equal to 19 years. In Japan, subjects must be aged greater than or equal to 20 years. In Singapore, subjects must be aged greater than or equal to 21 years.
* Histological evidence of NASH based on a central pathologist evaluation of the baseline liver biopsy. The baseline liver biopsy can be a historical biopsy obtained within 180 days prior to Visit 1.
* Histological evidence of fibrosis stage 2, 3 or 4 according to the NASH CRN classification based on a central pathologist evaluation of the baseline liver biopsy.
* Histological non-alcoholic fatty liver disease (NAFLD) activity score (NAS) greater than or equal to 4 for subjects with F2/F3 or greater than or equal to 3 for subjects with F4 based on a central pathologist evaluation of the baseline liver biopsy. All subjects must have a score of 1 or more in steatosis, lobular inflammation and hepatocyte ballooning.

Exclusion Criteria:

* Documented causes of chronic liver disease other than NAFLD.
* Positive HBsAg, positive anti-HIV, positive HCV RNA at screening (V2A) or any known presence of HCV RNA or HBsAg within 2 years of screening (V2A).
* Presence or history of ascites more than grade 1, variceal bleeding, hepatic encephalopathy, spontaneous bacterial peritonitis or liver transplantation at V2A.
* For subjects with F4, presence or history of gastro-oesophageal varices more than or equal to grade 2 at V3. An oesophagogastroduodenoscopy performed no more than 52 weeks prior to V3 must be available at V3.
* Known or suspected excessive consumption of alcohol (more than 20 g/day for women or more than 30 g/day for men) or alcohol dependence (assessed by the Alcohol Use Disorders Identification Test (AUDIT questionnaire)).
* Treatment with vitamin E (at doses more than or equal to 800 IU/day) or pioglitazone or medications approved for the treatment of NASH which has not been at a stable dose in the opinion of the investigator in the period from 90 days prior to V2A. In addition, for subjects with a historical liver biopsy taken more than 90 days prior to V2A, treatment should be at a stable dose in the opinion of the investigator from time of biopsy until V2A.
* Treatment with GLP-1 RAs within 90 days prior to V2A. Subjects with a historical liver biopsy taken more than 90 days prior to V2A are excluded if they receive treatment with GLP-1 RAs from time of biopsy until V2A.
* Treatment with glucose-lowering agent(s) (other than GLP-1 RAs), lipid-lowering medication or weight loss medication not stable in the opinion of the investigator in the period from 90 days prior to V2A. In addition, for subjects with a historical liver biopsy taken more than 90 days prior to V2A, treatment should be at a stable dose in the opinion of the investigator from time of biopsy until V2A.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 698 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Improvement in liver fibrosis and no worsening of NASH (Yes/No) | From baseline (week 0) to week 52
  Count of subjects Improvement in fibrosis is defined as greater than or equal to 1 grade improvement on the NASH CRN fibrosis scale

SECONDARY OUTCOMES:
Resolution of steatohepatitis and no worsening of liver fibrosis (Yes/No) | From baseline (week 0) to week 52
  Count of subjects Resolution of steatohepatitis is defined as a NAS of 0-1 for inflammation, 0 for ballooning and any value for steatosis according to NASH CRN52. Fibrosis is graded on the NASH CRN (Non-Alcoholic Steatohepatitis Clinical Research Network) fibrosis scale from 0 to 4.
Improvement in steatohepatitis with at least a 2-point reduction in NAS and no worsening of fibrosis (Yes/No) | From baseline (week 0) to week 52
  Count of subjects The 2-point reduction must include at least a 1-point reduction in either lobular inflammation or hepatocellular ballooning.
Change in histology-assessed liver collagen proportionate area | From baseline (week 0) to week 52
  Ratio to baseline
Resolution of steatohepatitis and improvement in liver fibrosis (Yes/No) | From baseline (week 0) to week 52
  Count of subjects Resolution of steatohepatitis is defined as an NAS score of 0-1 for inflammation, 0 for ballooning and any value for steatosis (according to NASH CRN).
  Improvement in fibrosis is defined as greater than or equal to 1 grade improvement on the NASH CRN fibrosis scale
Improvement in liver fibrosis (Yes/No) | From baseline (week 0) to week 52
  Count of subjects Improvement in fibrosis is defined as greater than or equal to 1 grade improvement on the NASH CRN fibrosis scale
Progression of liver fibrosis (Yes/No) | From baseline (week 0) to week 52
  Count of subjects For subjects with fibrosis stage 2 or 3 at baseline
Worsening in steatohepatitis (Yes/No) | From baseline (week 0) to week 52
  Count of subjects Worsening in steatohepatitis is defined as increase in NAS score for ballooning, inflammation or steatosis
Improvement in ballooning (Yes/No) | From baseline (week 0) to week 52
  Count of subjects
Improvement in inflammation (Yes/No) | From baseline (week 0) to week 52
  Count of subjects
Improvement in steatosis (Yes/No) | From baseline (week 0) to week 52
  Count of subjects
Change in ALT (alanine aminotransferase) | From baseline (week 0) to week 52
  Ratio to baseline
Change in AST (aspartate aminotransferase) | From baseline (week 0) to week 52
  Ratio to baseline
Change in inflammation assessed by HsCRP (high sensitivity C-reactive protein) | From baseline (week 0) to week 52
  Ratio to baseline
Change in ELF (Enhanced Liver Fibrosis) score | From baseline (week 0) to week 52
  Logarithm
Change in HbA1c. For subjects with type 2 diabetes | From baseline (week 0) to week 52
  %-points (absolute change)
Change in triglycerides | From baseline (week 0) to week 52
  Ratio to baseline
Change in free fatty acids | From baseline (week 0) to week 52
  Ratio to baseline
Change in LDL (low density lipoprotein) cholesterol | From baseline (week 0) to week 52
  Ratio to baseline
Change in HDL (high density lipoprotein) cholesterol | From baseline (week 0) to week 52
  Ratio to baseline
Relative change in body weight | From baseline (week 0) to week 52
  Percentage
Change in SF-36 (36-item Short Form Survey) bodily pain | From baseline (week 0) to week 52
  Points
Change in NASH-CHECK (patient-reported outcome measure for non-alcoholic steatohepatitis)pain | From baseline (week 0) to week 52
  Points
Change in PROMIS (Patient-Reported Outcomes Measurement Information System) Fatigue score | From baseline (week 0) to week 52
  Points
Number of treatment emergent adverse events (TEAEs) | From baseline (week 0) to week 59
  Count

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (254):
- United States (70):
  - North AL Health Res, LLC, Huntsville, Alabama
  - The Institute for Liver Health, Chandler, Arizona
  - Inst-Liver Hlth dba AZ Liver H, Peoria, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Hope Clinical Research, Canoga Park, California
  - UCSD NAFLD Research Center, La Jolla, California
  - OM Research LLC, Lancaster, California
  - Digestive Hlth Res of SoCa, Long Beach, California
  - Stanford Medicine, Redwood City, California
  - UC Davis Hlth -Midtwn Ambu Cen, Sacramento, California
  - Peak Gastro Assoc-Col Springs, Colorado Springs, Colorado
  - Hartford Hsptl_Hartford, Hartford, Connecticut
  - Integrity Clinical Research, LLC, Doral, Florida
  - Miguel Rebollar PA, Hialeah, Florida
  - Nature Coast Clinical Research_Inverness, Inverness, Florida
  - UF Hlth Jacksonville, Jacksonville, Florida
  - Florida Research Institute, LLC, Lakewood Rch, Florida
  - ClinCloud,LLC, Maitland, Florida
  - Optimus U, Corp, Miami, Florida
  - Univ of Miami/Schiff Ctr, Miami, Florida
  - Covenant Metabolic Specialists LLC, University Park, Florida
  - ClinCloud, LLC, Viera E., Florida
  - Florida Medical Clinic Orlando Health, Zephyrhills, Florida
  - Florida Medical Clinic, LLC, Zephyrhills, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Gastroenterology Assoc_ CGA, Macon, Georgia
  - Gastroint Spec of Georgia, Marietta, Georgia
  - EBGS Clinical Research Center, LLC, Snellville, Georgia
  - Grand Teton Gastroenterology, Idaho Falls, Idaho
  - Digestive Research Alliance of Michiana, South Bend, Indiana
  - University Of Kansas Hospital, Kansas City, Kansas
  - Kansas Medical Clinic, PA, Topeka, Kansas
  - Tandem Clinical Research - Houma, Houma, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Tandem Clinical Research - Metairie, Metairie, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Mercy Medical Center, GI Research, Baltimore, Maryland
  - Walter Reed Nat Mil Md Ctr, Bethesda, Maryland
  - Henry Ford Hospital_Detroit, Detroit, Michigan
  - Kansas City Research Institute, Kansas City, Missouri
  - Univ of Nebraska Medical CTR, Omaha, Nebraska
  - AIG Digestive Disease Research, Florham Park, New Jersey
  - NYU Grossman School of Med, New York, New York
  - Weill Cornell Med Coll-NYPH, New York, New York
  - Univ Hosp Cleveland Med Ctr, Cleveland, Ohio
  - Ohio State Univ Wexner Med Ctr, Columbus, Ohio
  - DSI Research,LLC, Springboro, Ohio
  - Geisinger Clinic, Danville, Pennsylvania
  - Pennsylvania State University, Hershey, Pennsylvania
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC Center for Liver Diseases, Pittsburgh, Pennsylvania
  - UPMC_Center for Liver Care, Pittsburgh, Pennsylvania
  - Digestive Health Res-TSMC, Hermitage, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Texas Clin Res Inst, LLC, Arlington, Texas
  - Liver Ins@ Mthdist DTX Med Cen, Dallas, Texas
  - Centex Studies, Inc., Houston, Texas
  - Amir Ali Hassan, MD, PA, Houston, Texas
  - Texas Diabetes &Endocrinology, Round Rock, Texas
  - Amer. Rrsch Corp-TX Liver Inst, San Antonio, Texas
  - Olympus Clinical Research, Sugar Land, Texas
  - Impact Research, Waco, Texas
  - Digestive Hlth Res of N Texas, Wichita Falls, Texas
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Bon Secours Richmond Community Hospital LLC, Richmond, Virginia
  - Gastroent Consult of SW VA, Roanoke, Virginia
  - Swedish med ctr org trans-lvr ctr, Seattle, Washington
  - Liver Institute NW, Seattle, Washington
- Australia (10):
  - Genesis Research Services, Broadmeadow, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital - Hepatology- 5E291, Adelaide, South Australia
  - Monash Health Department of Gastroenterology, Clayton, Victoria
  - St Vincent's Hospital (Melbourne), Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Centre - Gastroenterology, Melbourne, Victoria
  - Fiona Stanley Hospital - Hepatology, Murdoch, Western Australia
- Belgium (4):
  - CUB Hôpital Erasme_Brussels_0, Brussels
  - Cliniques Universitaires Saint-Luc - Serv. Hépato-gastroentérology, Brussels
  - UZA, Edegem
  - UZ Gent - Department Gastro-enterology, Ghent
- Bulgaria (8):
  - MHAT - UniHospital OOD, Panagyurishte
  - MHAT Med Line Clinic, Plovdiv
  - "Acibadem City Clinic UMHAT Tokuda", Sofia
  - DCC Aleksandrovska EOOD, Sofia
  - UMHAT "Sv. Ivan Rilski", Clinic of Gastroenterology, Sofia
  - Medical Center Vertebra OOD, Sofia
  - "UMHAT "Tsaritsa Yoanna-ISUL"" EAD, Gastroenterology clinic, Sofia
  - "DCC XX - Sofia" EOOD, Sofia
- Canada (7):
  - University of Calgary Liver Unit-(HMRC), Calgary, Alberta
  - GI Research Inst Foundation, Vancouver, British Columbia
  - QE II Health Sciences Centre, Halifax, Nova Scotia
  - LMC Manna Research Inc. (London), London, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Ctr de Med Metab de Lanaudiere, Terrebonne, Quebec
- Czechia (3):
  - Krajská nemocice Liberec, a.s, Liberec
  - Fakultni nemocnice Plzen - Lochotin, Pilsen
  - Vseobecna Fakultni nemocnice v Praze, Prague
- Denmark (3):
  - Hvidovre Hospital - Gastroenheden, Hvidovre
  - Abdominal Center K, Research Unit, København NV
  - Odense University Hospital, Odense C
- France (8):
  - Centre Hospitalier Universitaire D'Angers-1, Angers
  - Ap-Hp-Hopital Beaujon, Clichy
  - Centre Hospitalier Universitaire de Lille-Hopital Claude Huriez, Lille
  - Hospices Civils de Lyon-Hopital de La Croix Rousse, Lyon
  - Centre Hospitalier Universitaire de Nice-Hopital de L'Archet 2, Nice
  - Aphp-Hopital La Pitie Salpetriere-4, Paris
  - Centre Hospitalier Universitaire de Nantes-Hopital Nord Laennec-1, Saint-Herblain
  - Centre de Recherche Clinique Portes Du Sud, Vénissieux
- Germany (7):
  - Klinik für Endokrinologie, Diabetologie und Stoffwechsel, Essen
  - Uniklinik Schleswig-Holstein - Medizinischen Klinik I am Campus Lübeck, Lübeck
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsmedizin der JGU Mainz - Hepatologie, Mainz
  - Uniklinik Tübingen - Innere Medizin I, Tübingen
  - Universitätsklinikum Würzburg - Zentrum für Innere Medizin (ZIM), Würzburg
  - Universitätsklinikum Würzburg, ZIM, Würzburg
- Greece (5):
  - Gen Hospital of Athens Ippokrateio,B' Uni Clinic of Inte Med, Athens
  - Gen Hospital of Athens Laiko,1st Dpt. of Propaedeutic Inter, Athens
  - General Hospital of Athens "LAIKO", Goudi, Athens
  - "AHEPA" University Hospital of Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki "Ippokrateio", Thessaloniki
- India (18):
  - Yashoda Hospital, Secunderabad, Andhra Pradesh
  - Surat Institute of Digestive Science, Surat, Gujarat
  - BAPS Pramukh Swami Hospital, Surat, Gujarat
  - Medanta - The Medicity Multi-Speciality Hospital, Gurugram, Gurugram, Haryana
  - Kasturba Medical College Hospitals (KMC Hospitals), Mangalore, Mangalore, Karnataka
  - KLES & Prabhakar Kore Hospital and Research Centre, Belagavi, Karnatka
  - Gleneagles Hospital, Super-speciality and Transplant Centre, Parel, Mumbai, Maharashtra
  - Seth GS medical college and KEM Hospital, Mumbai, Maharashtra
  - Midas Multispeciality Hospital, Nagpur, Maharashtra
  - Institute of liver and Biliary Sciences, Ghitorni, New Delhi
  - All India Institute of medical Sciences, New Dehli, New Delhi
  - Fortis Heart Institute and Multispeciality Hospital, Chandigarh,, Punjab
  - Post Graduate Institute of Medical Education & Research_Chandigarh, Chandigarh, Punjab
  - Dayanand Medical College & Hospital, Ludhiana, Punjab
  - S.R.Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - SMS Medical College & Hospital, Jaipur, Rajasthan
  - Osmania General Hospital, Hyderabad, Telangana
  - Dr P V Rao - Diabetes Research Centre, Hyderabad, Telangana
- Italy (8):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona
  - Azienda Socio Sanitaria Territoriale (ASST) Papa Giovanni XXIII, Bergamo
  - Azieda Ospedaliero-Universitaria, Policlinico S. Orsola-Malp, Bologna
  - AOU Careggi Padiglione 16 San Luca, 3° piano, Florence
  - Azienda Ospedaliera di Padova Clin.Med.3, Padua
  - AOU Pisana Stabilimento di Cisanello EDIFICIO 6, Piano 5, Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli IRCS, Roma
  - Policlinico Università Campus Biomedico di Roma, Rome
- Japan (17):
  - Chiba University Hospital_Chiba-shi, Chiba, Chiba-shi, Chiba
  - Fukui-ken Saiseikai Hospital, Internal Medicine, Fukui-shi, Fukui
  - Hamamatsu University Hospital, Hamamatsu-shi, Shizuoka
  - JA Hiroshima General Hospital_Gastroenterology and Hepatology, Hatsukaichi-shi, Hiroshima
  - University Hospital Kyoto Prefectual University of Medicine, Kamigyo-ku, Kyoto
  - St. Marianna University School of Medicine Hospital, Kawasaki-shi, Kanagawa
  - Kumamoto Shinto General Hospital_Liver・Gastroenterology, Kumamoto-shi, Kumamoto
  - Toranomon Hospital, Hepatology, Minato-ku, Tokyo
  - Kawasaki Medical School General Medical Center_Internal Medicine, Okayama-shi, Okayama
  - Saga University Hospital_Liver Center, Saga-shi, Saga
  - Sendai Kousei Hospital, Sendai-shi, Miyagi
  - Saiseikai Suita Hospital, Gastroenterology, Suita-shi, Osaka
  - Ehime University Hospital_Department of Gastro.& Metabo., Toon-shi, Ehime
  - Ehime University Hospital, Toon-shi, Ehime
  - Saiseikai Wakayama Hospital_Gastroenterology, Wakayama-shi, Wakayama
  - Saiseikai Wakayama Hospital, Wakayama-shi, Wakayama
  - Yokohama City University Hospital, Gastrointestinal Medicine, Yokohama-shi, Kanagawa
- Malaysia (3):
  - Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Selayang, Batu Caves
- Poland (11):
  - ID Clinic Arkadiusz Pisula, Myslowice, Lesser Poland Voivodeship
  - Spolka Lekarzy Intercor Sp. z o.o., Bydgoszcz
  - Clinical Medical Research Korfantego - Ambulatoryjna Opieka, Katowice
  - Uniwersyteckie Centrum Kliniczne im. Prof. K. Gibińskiego Śl, Katowice
  - "LANDA" Katarzyna Agata Landa, Krakow
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Centrum Medyczne Medyk Sp. z o.o., Rzeszów
  - EMC Instytut Medyczny S.A., Wroclaw
  - Centrum Badan Klinicznych, Wroclaw
  - FutureMeds Sp. z o.o., Wroclaw
  - Velocity Nova Sp. z o.o., Staszów, Świętokrzyskie Voivodeship
- Portugal (3):
  - Unidade Local De Saude De Matosinhos E.P.E., Senhora Da Hora, Matosinhos, Matosinhos
  - Unidade Local De Saude De Santa Maria E.P.E., Lisbon
  - Hospital Luz Arrabida, S.A., Vila Nova de Gaia
- FDI Clinical Research, San Juan, Puerto Rico
- Russia (32):
  - Volosevich First City Clinical Hospital, Arkhangelsk
  - City Hospital #5, Barnaul
  - Limited Liability Company "Alliance Biomedical Ural Group", Izhevsk
  - Kazan Federal University, Kazan'
  - LLC "Clinic of Aesthetic Medicine & Laser Technologies", Kazan'
  - Limited Liability Company "Polyclinica № 1", Moscow
  - Friendship University of Russia, Moscow
  - FSBI 'I.I. Dedov National Medical Research Center of Endocrinology' of the MH of Russia, Moscow
  - Setchenov First Moscow State Medical University, Moscow
  - PHI "Central Clinical Hospital RZD- Medicine", Moscow
  - Pirogov Russian National Research Medical University MoH, Moscow
  - LLC RC Medical, Novosibirsk
  - RIIPM - branch of ICG SB of RAS, Novosibirsk
  - Limited Law Company "Healthy Family" Medicine Center", Novosibirsk
  - LLC "Clinical diagnostic center Ultramed", Omsk
  - BHI of Omsk Region "City Hospital № 3", Omsk
  - Penza Regional Clinical Hospital named after N.N. Burdenko, Penza
  - Joint Stock Company "Polyclinic Complex", Saint Petersburg
  - SPb SBHI City Outpatient clinic #109, Saint Petersburg
  - Limited Liability Company "Clinic" MEDINEF ", Saint Petersburg
  - Limited Liability Company "Energiya Zdoroviya", Saint Petersburg
  - X Seven Clinical Research Limited Liability Company, Saint Petersburg
  - SPb SBHI City polyclinic #117, Saint Petersburg
  - North-Western State Medical Univer. based on Med-Prof Center, Saint Petersburg
  - Medical Research Institute LLC, Saint Petersburg
  - Limited Liability Company "Research Center Eco-safety", Saint Petersburg
  - Private medical institution "Euromedservice", Saint Petersburg
  - Consultative & Diagnostic Center with a Outpatient Hospital, Saint Petersburg
  - Siberian State Medical University, Tomsk
  - Ulianovsk Regional Clinical Hospital, Ulyanovsk
  - Joint Stock Company "Medical technologies", Yekaterinburg
  - Polyclinic #2 in Yoshkar-Ola, Yoshkar-Ola
- Singapore (4):
  - National University Hospital_Tahir Building, Singapore
  - National University Hospital_TBD, Singapore
  - Singapore General Hospital, Singapore
  - Changi General Hospital, Singapore
- South Korea (10):
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Kyungpook National University Hospital, Daegu
  - Yeungnam Univ. Medical Center, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Wonju Severance Christian Hospital, Gangwon-do
  - SoonChunHyang University Hospital Bucheon, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Chung-Ang University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (6):
  - Complejo Hospitalario de Pontevedra - Hospital de Montecelo, Pontevedra, Galicia
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Virgen del Rocío, Seville
  - Hospital Clínico de Valladolid, Valladolid
- Taiwan (4):
  - Ditmanson Medical Foundation Chia-Yi Christian Hospital, Chiayi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital_main, Taipei
- Turkey (Türkiye) (9):
  - Hacettepe Universitesi Tıp Fakültesi- Gastroenteroloji, Ankara
  - Gazi University Medical Faculty, Ankara
  - Gaziantep Üniversitesi Hastanesi, Gaziantep
  - Bezmialem Vakıf Üniversitesi Hastanesi-Gastroenteroloji, Istanbul
  - Cerrahpasa Kardiyoloji Enstitüsü, Istanbul
  - Marmara Univ. Pendik Gastroenterology, Istanbul
  - Kocaeli Universitesi Tıp Fakültesi Gastroenteroloji ve Hepat, Kocaeli
  - Recep Tayyip Erdoğan Üniversitesi EAH-Endokrinoloji, Rize
  - Adana Şehir Eğitim ve Araştırma Hastanesi, Yüreğir/Adana
- United Kingdom (3):
  - Queen Elizabeth Hospital, Birmingham, Birmingham
  - Royal Devon & Exeter NHS Foundation Trust, Exeter
  - Imperial College London, London

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com